CLINICAL TRIAL: NCT01094431
Title: Infectious Disease Etiologies of Uncomplicated Febrile Illness in Children <5 Years of Age in Rural Zanzibar
Brief Title: Etiology of Uncomplicated Fever in Children <5 in Rural Zanzibar
Acronym: RDTNEG
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Zanzibar Malaria Control Programme (Other Government); World Health Organization (Other); Göteborg University (Other); Queen Silvia Children's Hospital, Gothenburg, Sweden (Other)
Responsible Party: Principal Investigator, Anders Björkman, Professor, Karolinska University Hospital
Other Study IDs: Fever 2010
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Fever; Infectious Disease
Keywords: Fever; Etiology; Children under five years of age; IMCI
MeSH Terms: conditions — Fever; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — Urine collected in deep ager Frozen Nasopharyngeal secretions
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to study the most common etiologies of uncomplicated fever diseases among children under five years of age in rural Zanzibar.

DETAILED DESCRIPTION:
During the last 6 years Zanzibar has undergone a dramatic change in malaria epidemiology and burden of disease, with a marked decline of Plasmodium falciparum malaria among febrile children from approximately 30% to 1% or below and a reduction of crude child mortality of 50%. Millions of children in Africa die of neonatal disorders, acute respiratory tract infections (ARI), diarrhea, malaria, measles, HIV and malnutrition. A majority of these illnesses are also a common cause of febrile illness in out-patient departments. However, most of the few fever studies made in Africa are hospital based Very few studies on etiology of childhood febrile disease have been conducted on first level health facilities in the least developed countries in Africa. This study will therefore focus on children between 2 months to 5 years of age that have been diagnosed with a negative rapid diagnostic test (RDT) for malaria and their causes of fever at the first referral level in out-patient clinics in Zanzibar.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 2-59 months of age with confirmed fever, with a measured axillary temperature of ≥37.5˚C, or history of fever within the preceding 24 hours.
* Presenting at the health facility from 8.00 to 16.00 Monday to Friday.
* Informed consent.
* Able and willing to complete stipulated follow-up.

Exclusion Criteria:

* Decision by the clinician to refer the patient to another health facility than the PHCC where the study is conducted.
* Symptoms/ signs of severe disease that requires immediate referral from the PHCC as defined by the clinicians. These symptoms/signs of severe disease are according to the IMCI guidelines.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Kivunge Primary Health Care Center (PHCC) in North A District in Zanzibar
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
relative frequency of febrile diseases etiology | Five months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, Professor, Principal Investigator — Karolinska University Hopsital; Magnus Lindh, Professor, Principal Investigator — Sahlgrenska University Hospital; Mwinyi Msellem, MSc, Principal Investigator — Zanzibar Malaria Control Programme; Abdullah S. Ali, Manager, Principal Investigator — Zanzibar Malaria Control Programme; Birger Trollfors, Professor, Principal Investigator — Sahlgrenska University Hospital; Andreas Mårtensson, MD, PhD,, Principal Investigator — Karolinska University Hospital; Kristina Elfving, M.D., Principal Investigator — Sahlgrenska University Hospital; Deler Shakely, M.D., Principal Investigator — Karolinska University Hopsital
Locations (1):
- Facility: Primary health care center (PHCC), Kivunge, North A district, Zanzibar, Kivunge, Zanzibar, Tanzania

REFERENCES:
- [Derived] Elfving K, Stromberg LG, Geravandi S, Andersson M, Bachelard M, Msellem M, Shakely D, Trollfors B, Norden R, Martensson A, Bjorkman A, Lindh M. Pneumococcal concentration and serotype distribution in preschool children with radiologically confirmed pneumonia compared to healthy controls prior to introduction of pneumococcal vaccination in Zanzibar: an observational study. BMC Infect Dis. 2022 Dec 10;22(1):925. doi: 10.1186/s12879-022-07902-5. PMID 36496395